CLINICAL TRIAL: NCT05476042
Title: The Effect of Local Erythropoietin 3000 and 6000 Units on the Treatment of Conjunctival and Scleral Avascular Lesions: A Multicenter Clinical Trial
Brief Title: The Effect of Erythropoietin in the Treatment of Scleral Necrosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14015
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Conjunctival and Scleral Avascular Lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescribe Erythropoieti (Active Comparator)
  Interventions: Drug: Erythropoietin prescription
- Prescribe placebo (Placebo Comparator)
  Interventions: Drug: Prescription of placebo

INTERVENTIONS:
Drug: Prescription of placebo — Normal saline
  Arms: Prescribe placebo
Drug: Erythropoietin prescription — Erythropoietin 3000 units in normal saline
  Arms: Prescribe Erythropoieti
Drug: Erythropoietin prescription — Erythropoietin 6000 units in normal saline
  Arms: Prescribe Erythropoieti

SUMMARY:
Patients with acute avascular lesions of the conjunctiva and sclera will be included in the study. Patients will undergo a complete eye examination including a slit lamp, intraocular pressure measurement, and fundoscopy with dilated pupil. At the same time, laboratory examination including measurement of fasting blood sugar (FBS) level, complete blood count (CBC) and systemic blood pressure will be performed. Patients will be randomly divided into three groups. The groups will receive sham drops (normal saline), erythropoietin 3000 units in normal saline, and erythropoietin 6000 units in normal saline every 6 hours respectively. Meanwhile, all patients will receive the usual treatments based on the cause of scleral necrosis.

Eye examinations will be done daily in the first week, every other day in the second week, and then twice a week until the complete recovery of avascular lesions. In each examination, with fluorescein staining, the size of the conjunctival epithelial defect will be determined. Also, the dimensions of the avascular area of the sclera will be determined. Other examinations include measurement of visual acuity and intraocular pressure, and the patient will be evaluated in terms of iris and retinal neovascularization. The photoslit lamp will be done before starting the study and then every week.

Complete healing of the lesion is defined by complete vascularization and epithelization of the ischemia site. After the complete recovery of conjunctival and scleral necrosis, the erythropoietin drop will be stopped and the examinations including blood pressure measurement, CBC, diff and FBS will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute conjunctival and scleral avascular lesions resulting from ocular surgery (such as pterygium resection, glaucoma, strabismus, vitreous and retinal surgery), chemical and thermal burns, and collagen-vascular disease.

Exclusion Criteria:

* a history of ocular surface tumors
* a history of tumors in any part of the body
* iris and retinal neovascularization for any reason
* proliferative diabetic retinopathy
* and systemic hypertension
* if the sclera is severely thinned and the risk of perforation of the globe is imminent, the patient is excluded from the study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-14 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The size of the conjunctival epithelial defect | 1 week
  Caliper

SECONDARY OUTCOMES:
The rate of angiogenesis at the site of the epithelial defect | 1 week
  Caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research center, Tehran, Iran